CLINICAL TRIAL: NCT04217304
Title: SONOthrombolysis in Patients With an ST-segment Elevation Myocardial Infarction With fibrinoLYSIS (SONOSTEMI-LYSIS) Trial
Acronym: SONOSTEMILYSIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00093814
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — perflutren

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sonothrombolysis (Experimental): Diagnostic myocardial contrast echocardiography with ultrasound contrast agent 5% Definity® plus Sonothrombolysis
  Interventions: Drug: Definity® with High Mechanical Index Ultrasound
- Standard of Care (No Intervention): Diagnostic myocardial contrast echocardiography with ultrasound contrast agent 5% Definity®

INTERVENTIONS:
Drug: Definity® with High Mechanical Index Ultrasound — Sonothrombolysis; Echocardiographic imaging with intermittent diagnostic high mechanical index during an intravenous 5% Definity® infusion
  Arms: Sonothrombolysis

SUMMARY:
This study will assess the safety and feasibility of sonothrombolysis in the acute management of STEMI undergoing reperfusion therapy with systemic fibrinolysis as part of a pharmacoinvasive approach

DETAILED DESCRIPTION:
This study is an open label, single-centre, randomized investigation of sonothrombolysis in 60 adult patients presenting with STEMI within 6 hours of the onset of clinical symptoms and receiving perfusion therapy with fibrinolysis as part of a pharmacoinvasive strategy.

Patients will be randomized 2:1 to either adjunct treatment with sonothrombolysis or standard therapy alone according to the current American College of Cardiology/American Heart Association (ACC/AHA) or European Society of Cardiology (ESC) STEMI and PCI guidelines. All patients will receive serial echocardiography assessments during and after reperfusion with the final ECHO assessment at 90 days (+/- 7d) post reperfusion. Patient outcomes (medical records review) will be followed for 1 year after reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with STEMI within 6 hours of symptom onset and:

  1. Are expected to receive reperfusion therapy with fibrinolysis
  2. Have a high-risk STEMI ECG as defined as:

     * >2mm ST-segment elevation in 2 anterior or lateral leads; or
     * >2mm ST-segment elevation in 2 inferior leads coupled with ST-segment depression in 2 contiguous anterior leads for a total ST-segment deviation of >4mm
  3. Age >30 years
  4. Adequate apical and/or parasternal images by echocardiography

Exclusion Criteria:

* 1. Isolated inferior STEMI without anterior ST-segment depression 2. Previous coronary bypass surgery 3. Cardiogenic shock 4. Known or suspected hypersensitivity to ultrasound contrast agent used for the study 5. Life expectancy of less than two months or terminally ill 6. Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors, anticoagulants, or aspirin 7. Known large right to left intracardiac shunts 8. Patient received another investigational medication or treatment within 30 days prior to presentation with STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete ST-Segment Resolution | 90 minutes post TNK administration
  ST-segment recovery as assessed by complete ST-segment resolution (>50%)

SECONDARY OUTCOMES:
Frequency of rescue/urgent PCI | approximately 3-24 hours post TNK administration
  Frequency of rescue/urgent PCI following the administration of fibrinolysis.
ST-segment resolution (>50%) | approximately 30 minutes post TNK administration
  ST-segment resolution (>50%) following a pharmacoinvasive approach at ~30 minutes post PCI as assessed by the worst lead on electrocardiogram
ST-segment resolution (continuous) | approximately 30 minutes post TNK administration
  ST-segment resolution (continuous) following a pharmacoinvasive approach at ~30 minutes post PCI as assessed by the worst lead on electrocardiogram
Left ventricular ejection fraction | Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
  Left ventricular ejection fraction by ECHO (Simpson method) assessed on Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
Wall motion score index (WMSI) | Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
  Wall motion score index (WMSI) by ECHO assessed on Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
  Each of the 17 LV segments is classified as:
  1 normal 2.hypokinetic 3.akinetic 4.dyskinetic The WMS index is the sum of the scores divided by the number of segments. Usually 17, but if a segment cannot be classified, the sum is divided by the number of readable segments.
  Minimum value is 1 : all segments are normal - best outcome Maximum value is 4: all segments are dyskinetic - worst outcome
Microvascular perfusion score index (MPSI) | Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
  Microvascular perfusion score index (MPSI) by ECHO assessed on Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction
  Each of the 17 LV segments is classified as:
  1. normal, contrast replenishment within 4 seconds
  2. mildly reduced, contrast replenishment takes longer than 4 seconds
  3. no contrast replenishment over 10 seconds
  The MPSI index is the sum of the scores divided by the number of segments. Usually 17, but if a segment cannot be classified, then the sum is divided by the number of readable segments
  Minimum value is 1 : all segments are normal - best outcome Maximum value is 3: all segments are not perfused - worst outcome
Global Longitudinal Strain (GLS) | Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction.
  Global Longitudinal Strain (GLS) by ECHO assessed on Day 1 (pre reperfusion), Day 3 +/-2d (hospital discharge), and Day 90 +/-2d after infarction
  GLS is measured using speckle tracking imaging (Epiq, Philips). The scale is - % which means percentage of longitudinal shortening of myocardial segments. Similar to the WMSI, GLS is calculated by dividing the sum of the longitudinal strain measurements in the myocardial segments segments by the number of segments which can be assessed by speckle tracking (18 when all segments in all 3 apical views can be analysed.
  The lower the absolute strain value the worse the LV function.
QRS Score | Day 3 +/-2d (hospital discharge)
  Selvester QRS Scoring System, assessed on Day 3 +/-2d (hospital discharge) ECG. Minimum score 0, Maximum score 32. Higher score indicates worse outcome.

OTHER OUTCOMES:
Composite of death/shock, heart failure/new myocardial infarction in hospital | Until hospital discharge, approximately 5 days
  Composite of death/shock, heart failure/new myocardial infarction in hospital
Composite of death/shock, heart failure/new myocardial infarction at 1-year | 1 year
  Composite of death/shock, heart failure/new myocardial infarction at 1-year
TIMI flow grade pre and post PCI on index angiogram | pre and post PCI on index angiogram, approximately 3-24 hours post TNK administration
  TIMI flow grade pre and post PCI on index angiogram

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No